CLINICAL TRIAL: NCT03086889
Title: Immersive Virtual Reality Based Training for Motor Function Rehabilitation of Upper Limbs After Subacute Stroke：Study Protocol of a Randomized Clinical Trial
Brief Title: Immersive Virtual Reality Based Training for Rehabilitation of Subacute Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trials were stopped after recruiting 60% of the planned sample after a median of 3 months follow-up and one interim analysis. The immersive virtual reality based training has proven to work.
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Song-he Jiang, Principal Investigator, Second Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KFYXK001
Record Dates: First submitted 2017-03-09; First posted 2017-03-22 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Immersion Virtual Reality Training ,Stroke, Upper Extremity, Randomized Controlled Trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group (Experimental): The intervention group will participate in immersion virtual reality based rehabilitation training for 3 weeks.
  Interventions: Other: immersion virtual reality (VR)-based rehabilitation
- The control group (Other): The control group will receive for traditional rehabilitation training for 3 weeks.
  Interventions: Other: traditional rehabilitation training

INTERVENTIONS:
Other: immersion virtual reality (VR)-based rehabilitation — Intervention group received VR-based rehabilitation,including Virtual kitchen and so on.The patients took part in the exercise program for 30 minutes each day, five times per week, for 3 weeks. All subjects received physiotherapy, which accounts for an average of 30 minutes of physiotherapy per day on tolerance.
  Arms: The intervention group
Other: traditional rehabilitation training — The traditional rehabilitation training included occupational therapy and physical therapy, patients took part in the traditional rehabilitation training for 60 minutes each day, five times per week, for 3 weeks.
  Arms: The control group

SUMMARY:
The investigators will conduct a single-blind, randomized controlled trial of 60 patients with subacute stroke. Patients will be randomly assigned into a control group and an intervention group. The intervention group will participate in immersion VR training for 3 weeks. The control group will receive for traditional rehabilitation training for 3 weeks. Then, the patients will be reevaluated to determine changes in upper extremity function, cognitive function, cortical and subcortical activation patterns, and performance of activities of daily living after the baseline assessment.

ELIGIBILITY:
Inclusion Criteria:

1. having had an ischemic stroke in the first time
2. age 30 to 80 years old
3. first stroke within 2 month
4. GCS score >8
5. the upper-limb function BrunnstromⅡ、Ⅲ

Exclusion Criteria:

1. hemorrhage or transient ischemic attack(TIA)
2. important organs such as heart, lung, liver, kidney function decline or failure
3. previous history of brain neurosurgery or epilepsy
4. had severe cognitive impairments or aphasia, which made the participants unable to understand the instructions given by the investigators
5. with claustrophobia and body with metal (such as metal teeth, etc.) are not suitable for to MRI scanning

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Arm Movement Ability at 3 months | Baseline and at 3 months
  The Fugl-Meyer Assessment

SECONDARY OUTCOMES:
Change from Baseline Activities of Daily Living (ADL) at 3 months | Baseline and at 3 months
  The Barthel index
Change from Baseline Cognitive Function at 3 months | Baseline and at 3 months
  the Korea-MiniMental Status Evaluation (K-MMSE)
Change from Baseline Cortical and Subcortical Activation Patterns at 3 months | Baseline and at 3 months
  Functional MRI (fMRI)

CONTACTS AND LOCATIONS:
Locations (1):
- Songhe Jiang, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Huang Q, Jiang X, Jin Y, Wu B, Vigotsky AD, Fan L, Gu P, Tu W, Huang L, Jiang S. Immersive virtual reality-based rehabilitation for subacute stroke: a randomized controlled trial. J Neurol. 2024 Mar;271(3):1256-1266. doi: 10.1007/s00415-023-12060-y. Epub 2023 Nov 10. PMID 37947856
- [Derived] Huang Q, Wu W, Chen X, Wu B, Wu L, Huang X, Jiang S, Huang L. Evaluating the effect and mechanism of upper limb motor function recovery induced by immersive virtual-reality-based rehabilitation for subacute stroke subjects: study protocol for a randomized controlled trial. Trials. 2019 Feb 6;20(1):104. doi: 10.1186/s13063-019-3177-y. PMID 30728055